CLINICAL TRIAL: NCT06798818
Title: Lung-cOnservative Liquid VEntilation for the Induction of Ultra-Rapid COOLing After Cardiac Arrest
Acronym: OverCool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ORIXHA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR23_0007; CIV-24-02-046114 (Other: EUDAMED)
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest; Post Cardiac Arrest Syndrome
Keywords: Cooling; Targeted Temperature Management; ROSC; Resuscitated Cardiac Arrest; Out of Hospital cardiac arrest; Therapeutic Hypothermia; liquid ventilation
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Vent2Cool device (Experimental): Vent2Cool is to be used to perform induction of Ultra-Rapid Therapeutic Hypothermia for the patients. The hypothermia maintenance and rewarming phases will be performed with an external TTM device as currently used in the investigation centres.
  Interventions: Device: Ultra-rapid therapeutic hypothermia induction by total liquid ventilation

INTERVENTIONS:
Device: Ultra-rapid therapeutic hypothermia induction by total liquid ventilation — Vent2Cool System is a targeted temperature management device used to induce ultra-rapid therapeutic hypothermia by total liquid ventilation.

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) affects over 356,000 individuals annually in the United States, with fewer than 10% surviving to hospital discharge, mirroring statistics from Europe. Post-cardiac arrest syndrome (PCAS), a condition causing multi-organ dysfunction, is a leading cause of mortality despite successful resuscitation efforts. Targeted temperature management (TTM) is recommended for comatose patients post-resuscitation to mitigate PCAS, but optimal temperature targets and cooling methods remain unclear. Experimental studies suggest that therapeutic hypothermia (32-34°C), induced rapidly after resuscitation, may provide significant clinical benefits.

Total liquid ventilation (TLV) with breathable liquids has been proposed to achieve ultra-rapid therapeutic hypothermia (URTH). This approach uses the lungs as a heat exchanger to achieve ultra-rapid cooling while maintaining normal gas exchange. It enables a reduction in core body temperature to the hypothermic range (33.0 ± 0.5°C) within 45 minutes in relevant experimental models.

The OverCool study is an open-label, single-arm, multi-centric pilot trial designed to evaluate the performance and safety of Vent2Cool, a medical device intended to induce ultra-rapid therapeutic hypothermia by TLV in resuscitated cardiac arrest patients. The primary objective is to demonstrate Vent2Cool's ability to achieve a target core temperature of 33.0 ± 0.5°C within 60 minutes from start of procedure in resuscitated patients admitted to the Intensive Care Unit following intra- or extra-hospital cardiac arrest. Secondary objectives include assessing procedural safety, cooling performance, feasibility in emergency settings, clinical outcomes, and the impact on biological markers.

DETAILED DESCRIPTION:
The "American Heart Association's 2022 Update" estimates that over 356,000 out-of-hospital cardiac arrests (OHCA) occur annually in the United States. These figures are consistant with data from European countries, where fewer than 10% of OHCA patients survive, despite 30% being successfully resuscitated before admission to intensive care units (ICU). The majority of these patients succumb to post-cardiac arrest syndrome (PCAS), a condition characterized by multi-organ failure.

To mitigate the severity of PCAS, current guidelines recommend continuous core temperature monitoring and active fever prevention through targeted temperature management (TTM) in patients who remain comatose following resuscitation from cardiac arrest. While TTM with a target temperature range of 32-36°C has been previously evaluated and applied in specific subpopulations, there is insufficient evidence to universally recommend one target temperature over another within this range. Conversely, experimental studies have demonstrated that the protective effects of therapeutic hypothermia (32-34°C) are strongly influenced by the rate of cooling initiated after resuscitation. These findings suggest that very early application of hypothermia may provide greater benefits compared to simply avoiding fever, emphasizing the importance of timely intervention.

In this context, Total Liquid Ventilation (TLV) with breathable liquids has been investigated in animal studies as a method to achieve ultra-rapid therapeutic hypothermia (URTH) following cardiac arrest. This innovative approach uses the lungs as a potent heat exchanger to achieve ultra-rapid cooling while preserving normal gas exchanges. TLV has demonstrated the capability to lower body core temperature from normothermia to the hypothermic range within 45 minutes, irrespective of body weight, in relevant experimental models. Furthermore, unlike earlier techniques of partial liquid ventilation, this method employs a lung-conservative liquid ventilation approach, which has been shown to be safe. The objective of the present OverCool study is to evaluate the performance and safety of the Vent2Cool device, designed to induce URTH by TLV safely following cardiac arrest.

Accordingly, OverCool is an open-label, single arm, non-comparative, multi-centric pilot study. The study primary objective is to demonstrate the ability of Vent2Cool to achieve a core body temperature of 33.0±0.5°C in less than 60 min after the start of the procedure in resuscitated patients admitted in the ICU after an intra- or extra-hospital cardiac arrest. The main secondary objectives are to demonstrate the safety of the procedure, the cooling performance, the ability to implement the procedure in the emergency setting of post-cardiac arrest management, the clinical outcomes and impact on biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Patient resuscitated after extra- or intra-hospital cardiac arrest, from presumed cardiac or asphyxial origin, regardless of the heart rate initially recorded.
* Age between 18 and 84 years old
* Time between collapse and return of spontaneous circulation (ROSC) < 60 min
* Presumption, at the time of inclusion, of a possibility of starting Vent2Cool within a period of less than 120 min after ROSC.
* Unconscious (GCS <8, not able to obey verbal commands after sustained ROSC)
* Patient affiliated with a social security system (If applicable)
* Consent of the member of patients' family or that of the trusted person if present and able to understand; otherwise certificate of emergency inclusion in compliance with applicable regulations.
* Vent2Cool must be connected to a standard cuffed ETT of 7.0 mm to 9.0 mm internal diameter for the procedure.

Exclusion Criteria:

* Conscious patient
* Patient Ideal Body Weight less than 40 kgs or more than 93 kgs
* Traumatic cardiac arrest, drowning, exsanguination, or sepsis
* Temperature at admission < 34.0°C
* Need for veno-arterial extracorporeal circulation (Extracorporeal membrane of oxygenation, ECMO) before return of spontaneous circulation (refractory cardiac arrest)
* One of the following signs at echocardiography at hospital admission:

  * Acute cor pulmonale, defined by right ventricular enlargement with interventricular septal deviation, associated with a Tricuspid Annular Plane Systolic Excursion (TAPSE) < 12 mm and need for vasopressor agents
  * Time-velocity integral of subaortic flow < 10 m/s
* Wrong positioning or damage of the endotracheal tube.
* Women under 50 years old (childbearing age) or for women of >50 years old, a positive pregnancy test (urinary) in case of pregnancy suspicion by the investigator. Possible breastfeeding during the study.
* Suspicion of intracranial bleeding
* History of severe Chronic Obstructive Pulmonary Disease (COPD) with long-term home oxygen therapy
* Acute respiratory pathology (pneumothorax, pleurisy, pneumonia, suspicion of contusion or intra-pulmonary hemorrhage following resuscitation)
* COVID-19 positive test in case of clinical suspicion and/or epidemic context
* Excessive mucus in the upper airways
* Patient presenting at least one of the following criteria in the mechanical ventilation parameters at inclusion:

  * PEEP > 8 cm H2O
  * Plateau pressure> 25 cmH2O
  * Driving pressure> 15cmH2O
* Patient with at least one of the following criteria at inclusion:

  * PaO2< 80 mmHg
  * PaO2 / FiO2< 150 mmHg
  * PaCO2> 48 mmHg

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of the Vent2Cool procedure (safe induction of ultra-rapid therapeutic hypothermia) | From start of Vent2Cool procedure to 60min after
  The primary end point is the success of the procedure. The success of the procedure is defined as the ability to reach a body core temperature (bladder temperature recommended) of 33.0±0.5°C and a safe return to conventional mechanical ventilation within less than one hour after Vent2Cool start. Start of the Vent2Cool procedure is defined as the opening of the Vent2Cool patient connector valve.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | At Day 28
  mRS will be evaluated at Day 28. The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symptoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.
Body Core Temperature | From start of Vent2Cool procedure to 37 hours after
  Core temperature (bladder recommended) at start of Vent2Cool procedure and for 36 h after the end of Vent2Cool procedure to include the maintenance and rewarming phases of TTM
Delay between the start of the Vent2Cool procedure and body core temperature of 33,5°C | During the Vent2Cool procedure
  Duration in minutes from start of the Vent2Cool procedure (i.e. opening of the Vent2Cool patient connector valve) to Body Core Temperature inferior or equal to 33,5 °C
Delay between return of spontaneous circulation (ROSC) and body core temperature of 33.5°C. | From ROSC to end of Vent2Cool procedure
  Duration in minutes from ROSC to body core temperature inferior or equal to 33,5 °C
PaO2 and PaCO2 | Inclusion, 10 min and 25 min after start of Vent2Cool procedure
  PaO2 and PaCO2 values from arterial blood gases sampled at inclusion and 10 and 25 minutes into the Vent2Cool procedure
Patient Vital status | Until Day 28
  Patient Vital status collected at ICU discharge and/or Hospital discharge (if before Day 28) and systematically at Day 28. In case of death : cause of death
Glasgow Outcome Score (GOS) | At Day 28
  The Glasgow Outcome Scale (GOS) is an ordinal scale used to assess functional outcomes of patients following brain injury.
  GOS includes five grades: 5, good recovery; 4, moderate disability; 3, severe disability; 2, persistent vegetative; and 1, death.

OTHER OUTCOMES:
Cooling Rate in body core temperature | During the Vent2Cool procedure
  Cooling rate is expressed in °C/h and calculated as follows: temperature at start of Vent2Cool procedure - 33.5°C / duration to achieve a core temperature of 33.5°C
Occurence of cooling overshoot | From start of Vent2Cool procedure to 60min after.
  Number and percentage of patients for whom the core temperature value is lower than 32°C and / or 30°C within 60 minutes after the start of the Vent2Cool procedure
Early termination of the Vent2Cool procedure by the clinician before reaching a core target temperature below 33±0.5°C (failure of cooling induction) | During the Vent2Cool procedure
modified Cardiac Arrest Hospital Prognosis (mCAHP) Score | At inclusion
  Value of the modified Cardiac Arrest Hospital Prognosis (mCAHP) Score. Scores of either <80; [80; 105[ or >105 predict of risk of poor outcomes of respectively at least 40%, at least 80% or at least 95%.
Prognostication according to the modified Cardiac Arrest Hospital Prognosis (mCAHP) score | At inclusion
  Number of patients for which the mCAHP score predicted a poor outcome with a risk of at least 40 % (mCAHP <80), at least 80% (mCAHP [80; 105[) or at least 95 % (mCAHP ≥ 105) vs. the total number of patients within each mRS category at Day 28.
Neurofilament light chain (NFL) | At inclusion, Day1 and Day3
Neuron Specific Enolase (NSE) | At inclusion, Day 1 and Day 3
Heart rate measured from the EKG or invasive blood pressure signal | At inclusion, 10 min and 25 min after start of Vent2Cool procedure
Systemic systolic and diastolic invasive blood pressure | At inclusion, 10 min and 25 min after start of Vent2Cool procedure
Presence of arrhythmia or unexpected electrocardiographic abnormality on EKG examination during Vent2Cool procedure | During the Vent2Cool procedure
Occurrence of an episode of major systemic hypotension (invasive or non-invasive measurement) with systolic blood pressure < 60 mmHg during Vent2Cool procedure | During the Vent2Cool procedure
Presence or absence of pleural collection of perfluorocarbon in the lungs on thoracic computed tomography examination in patients surviving on Day 28 after cardiac arrest. | Day 28
  The images of the CT scans will also be kept for possible later centralized analyses, if necessary.
Glasgow Coma Scale score | At inclusion, at Day 3 and at Day 28.
SOFA score | At Day 1 and Day 3
Percentage of patient with pulmonary infection | At Day 3
Oxygen desaturation based on SpO2 | During Vent2Cool procedure.
  Occurence of desaturation episodes defined as SpO2<75% on pulsed oxymeter lasting at least 5 minutes during Vent2Cool procedure.
Number and percentage of patients with severe hypercapnia | At inclusion, 10 min and 25 min after start of Vent2Cool procedure
  Severe hypercapnia defined as PaCO2>75 mmHg, in blood gases sampled at 10 and 25 minutes after start of Vent2Cool
Number and Percentage of patients with severe hyperoxemia | At inclusion, 10 min and 25 min after start of Vent2Cool procedure
  Severe hyperoxemia defined as PaO2>400 mmHg, in blood gases sampled at 10 and 25 minutes after start of Vent2Cool
Number and Percentage of patients with hypoxemia | At inclusion, 10 min and 25 min after start of Vent2Cool procedure
  Hypoxemia defined as PaO2 < 75 mmHg, in blood gases sampled at 10 and 25 minutes after start of Vent2Cool
Pupillometry examination | Day 1 to Day 3
  Presence of pupillary light reflex and Neurological pupil index (NPi) at Day 1, 2 and 3
Time of start of Vent2Cool procedure from the time of return of spontaneous circulation (ROSC) | From return of spontaneous circulation to start of Vent2Cool procedure
  Duration in minutes from ROSC to start of the Vent2Cool TLV procedure
Time of start of Vent2Cool procedure from the patient's admission to ICU | From patient admission to ICU to start of Vent2Cool procedure
Duration of the Vent2Cool procedure | From the start of the Vent2Cool procedure to the end of the procedure
  Time during which the patient is ventilated by Vent2Cool form start of Vent2Cool to end of TLV by lung draining procedure.
Vent2Cool performance parameters | During Vent2Cool procedure.
  based on device data recorded during the Vent2Cool procedure
Ventilatory parameters after Vent2Cool procedure | At 1h, 2h, 12h, 24h, 48h and 72h after the start of the Vent2Cool procedure
  Including measured values of:
  * positive end-expiratory pressure (PEEP),
  * end-inspiratory pause pressure (Plateau pressure),
  * driving pressure and static pulmonary compliance.
Hospital Care data | Until Day 28
  For patients discharged alive from hospital and / or alive at Day 28.
  * Number of days under mechanical ventilation
  * Number of days in intensive care unit
  * Number of days before hospital discharge, if applicable

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Cochin - Service de Medecine intensive et reanimation au 27 rue du Faubourg Saint-Jacques, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided